CLINICAL TRIAL: NCT00093626
Title: A Phase II Evaluation of BAY 43-9006 (Sorafenib, Nexavar®, NCI-Supplied Agent, NSC #724772) in the Treatment of Persistent or Recurrent Epithelial Ovarian or Primary Peritoneal Carcinoma
Brief Title: Sorafenib in Treating Patients With Persistent or Recurrent Ovarian Epithelial or Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02624; NCI-2012-02624 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000389246; GOG-0170F (Other: Gynecologic Oncology Group); GOG-0170F (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Primary Peritoneal Carcinoma; Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Sorafenib Tosylate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Sorafenib Tosylate — Given orally
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib

SUMMARY:
Sorafenib may stop the growth of tumor cells by stopping blood flow to the tumor and by blocking the enzymes necessary for their growth. This phase II trial is studying how well sorafenib works in treating patients with persistent or recurrent ovarian epithelial or peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of sorafenib in patients with persistent or recurrent ovarian epithelial or primary peritoneal carcinoma.

II. Determine 6-month progression-free survival of patients treated with this drug.

III. Determine the toxicity of this drug, in terms of frequency and severity of adverse events encountered, in these patients.

SECONDARY OBJECTIVES:

I. Determine the clinical response rate (partial and complete response) in patients treated with this drug.

II. Determine the duration of progression-free and overall survival of patients treated with this drug.

III. Correlate prognostic variables (platinum sensitivity, performance status, and histology [clear cell and mucinous type]) with response in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: Approximately 22-60 patients will be accrued for this study within 6-13 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian epithelial or primary peritoneal carcinoma

  * Persistent or recurrent disease
* Measurable or evaluable disease

  * Measurable disease is defined as at least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques (including palpation, plain x-ray, CT scan, or MRI) OR ≥ 10 mm by spiral CT scan
  * Evaluable disease is defined as at least 1 of the following:

    * CA 125 ≥ 2 times upper limit of normal (ULN)
    * Ascites and/or pleural effusion attributed to tumor
    * Solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST definition for target lesions
* Must have received 1 prior platinum-based chemotherapeutic regimen for primary disease, including carboplatin, cisplatin, or another organoplatinum compound

  * Initial treatment may have included high-dose therapy, consolidation, or extended therapy administered after surgical or non-surgical assessment
  * Platinum-resistant according to 1 of the following criteria:

    * Treatment-free interval of < 12 months after platinum therapy
    * Disease progression during platinum-based therapy
    * Persistent disease after a platinum-based regimen
* Ineligible for higher priority GOG protocol (e.g., any active phase III GOG protocol for the same patient population)
* No brain metastases
* Performance status - GOG 0-2 (for patients who received 1 prior treatment regimen)
* Performance status - GOG 0-1 (for patients who received 2 prior treatment regimens)
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No known bleeding diathesis
* Bilirubin ≤ 1.5 times ULN
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No uncontrolled hypertension
* Able to take oral medication
* No bowel obstruction or persistent vomiting
* No requirement for parenteral feedings
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study participation
* No sensory or motor neuropathy > grade 1
* No active or ongoing infection requiring antibiotics
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to sorafenib
* No serious chronic skin conditions (i.e., psoriasis or dermatitis) that would preclude study participation
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* At least 3 weeks since prior immunologic agents for the malignancy
* More than 4 weeks since prior mouse antibodies (for patients with evaluable disease only)
* No concurrent prophylactic growth factors (e.g., filgrastim [G-CSF])
* No concurrent prophylactic thrombopoietic agents except in the case of recurrent grade 4 thrombocytopenia
* No other concurrent biological agents for the primary tumor
* See Disease Characteristics
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior non-cytotoxic chemotherapy for persistent or recurrent disease
* No concurrent chemotherapy for the primary tumor
* At least 1 week since prior hormonal therapy for the malignancy
* No concurrent hormonal therapy for the primary tumor

  * Concurrent hormone replacement therapy allowed
* More than 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to > 25% of marrow-bearing areas
* No concurrent radiotherapy
* More than 4 weeks since prior surgery involving the peritoneum or pleura (for patients with evaluable disease only)
* Recovered from prior surgery
* At least 3 weeks since other prior therapy for the malignancy
* No more than 1 additional prior cytotoxic regimen for persistent or recurrent disease
* No prior sorafenib
* No prior anticancer treatment that would preclude study participation
* No concurrent therapeutic oral anticoagulation therapy (i.e., warfarin)

  * Concurrent prophylactic anticoagulation (i.e., low-dose warfarin) for central venous access devices allowed provided INR is < 1.5
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial agents or therapies for the malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2004-10; Primary Completion 2007-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of adverse events as assessed by CTCAE v3.0 | Up to 5 years
Progression-free survival | 6 months
  Will be evaluated using proportional hazards modeling and Fisher's exact test.

SECONDARY OUTCOMES:
Duration of overall survival | Up to 5 years
  Will be evaluated using proportional hazards modeling and Fisher's exact test.
Duration of progression-free survival | Up to 5 years
  Will be evaluated using proportional hazards modeling and Fisher's exact test.
Frequency of clinical response (complete and partial response) defined by RECIST criteria | Up to 5 years
Prognostic variables (platinum sensitivity, performance status, and cellular histology [clear cell or mucinous type]) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Matei, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States